CLINICAL TRIAL: NCT01098123
Title: Nutritional and Metabolic Context in Rowers
Brief Title: Metabolic Effects of Rowing Multi-races Events
Status: Completed | Type: Observational
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: F Desgorces, University Paris Descartes
Other Study IDs: 2006-A01070-57
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2006-02

CONDITIONS: Diet; Nutritional Status; Fatigue; Maximal Exercise
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diet counseling, nutritional index: Lightweight as athletes with weight limit
- nutritional index: Heavyweight athletes without weight limit

SUMMARY:
The aim of this study was to assess the relevance of NRI or athletes' NRI (ANRI) utilization to detect nutrition-related risks of failure in competition in the particular population of rowers.

In the morning, 60 to 90 minutes before the first race of a national level multi-races competition (three races for each subjects), body weight were measured and blood samples were collected with subjects at rest and in post-absorptive condition (last meal at least 2.5 hours before blood collection). Body weight was also recorded in the same conditions six weeks before the competition to calculate weight state (actual weight /usual weight ´ 100) and subjects were asked to identify the date of diet beginning. Body weight was measured using a floor scale (Mettler-Toledo floor scale, France), body mass index (BMI) was calculated from the ratio of weight (in kg) by height squared (in meters) and training volume (total duration of training in a week) was determined after discussion with athletes and coaches.

ELIGIBILITY:
Inclusion Criteria:

Competitors, volunteers

Exclusion Criteria:

non competitors

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Competitive athletes
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2006-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Infrared spectroscopy for serum albumin concentrations determinations | 30/05/2006

SECONDARY OUTCOMES:
Assessment of fatigue clinical signs | 25/04/06
  assessment of fatigue clinical signs by questionnary

CONTACTS AND LOCATIONS:
Overall Officials: François Desgorces, PhD, Principal Investigator — University Paris Descartes
Locations (1):
- INSEP, Paris, France

REFERENCES:
- [Background] Bouillanne O, Morineau G, Dupont C, Coulombel I, Vincent JP, Nicolis I, Benazeth S, Cynober L, Aussel C. Geriatric Nutritional Risk Index: a new index for evaluating at-risk elderly medical patients. Am J Clin Nutr. 2005 Oct;82(4):777-83. doi: 10.1093/ajcn/82.4.777. PMID 16210706